CLINICAL TRIAL: NCT01028898
Title: Screening and Identification of Abnormal Expression Proteins and miRNA From Colonic Mucosa of Patients With Irritable Bowel Syndrome.
Brief Title: Abnormal Expression Proteins, Mitochondrial DNA and miRNA of Irritable Bowel Syndrome
Acronym: IBS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: YANG Yun-sheng, ChinaPLAGH
Other Study IDs: IBS and metabolism
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2006-12

CONDITIONS: Irritable Bowel Syndrome; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Colonic Diseases; Colonic Diseases, Functional
Keywords: IBS; proteomics; fluorescent quantitation polymerase chain reaction; Western blot; immunohistochemistry staining (IHC); ATP content; micRNA
MeSH Terms: conditions — Irritable Bowel Syndrome; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Colonic Diseases; Colonic Diseases, Functional

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators enrolled IBS-D and IBS-C patients on the Rome III criteria and healthy volunteers as normal control group. Biopsies were taken from the cecum and sigmoid colon under direct vision. Five pieces were taken separately at each site. Four pieces were processed by cold saline water and frozen in liquid nitrogen immediately while the other one was fixed in formalin and then embedded in paraffin three days later.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In the investigators study, the investigators will focus on the screening of the related proteins and miRNA to IBS in order to reveal the possible clues or molecular mechanism for this disorder.

DETAILED DESCRIPTION:
For the proteomic procedures, Our study groups extracted proteins from the cecum and sigmoid colon samples and ran on the two-dimensional gel electrophoresis (2-DE). The proteins on 2-DE were visualized by the silver stain, and then gel maps were scanned and analyzed with the Image Master 2D Elite. The obvious abnormal protein spots were identified by the mass spectrometry. Western blot 、 immunohistochemistry 、 mRNA and miRNA were also performed for further verification of the proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms meeting Rome III criteria for diagnosis of IBS-C and IBS-D

Exclusion Criteria:

* Patients with organic illnesses or a history of major abdominal surgery
* Major psychotic episode, mental retardation or dementia
* Pregnant women and lactational women
* Postinfectious IBS, PI-IBS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IBS patients (IBS-D and IBS-C)and healthy control
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-08 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: YANG Yun-sheng, MD, Study Chair — Chinese PLA General Hospital; ZHANG Chun-yan, doctor, Principal Investigator — Chinese PLA General Hospital; WANG Weifeng, doctor, Principal Investigator — Chinese PLA General Hospital; YAO XIN, DOCTOR, Principal Investigator — Chinese PLA General Hospital; PENG LIHUA, DOCTOR, Principal Investigator — Chinese PLA General Hospital; YU YUANZI, DOCTOR, Principal Investigator — Chinese PLA General Hospital

REFERENCES:
- [Derived] Wang WF, Li X, Guo MZ, Chen JD, Yang YS, Peng LH, Wang YH, Zhang CY, Li HH. Mitochondrial ATP 6 and 8 polymorphisms in irritable bowel syndrome with diarrhea. World J Gastroenterol. 2013 Jun 28;19(24):3847-53. doi: 10.3748/wjg.v19.i24.3847. PMID 23840124